CLINICAL TRIAL: NCT01595412
Title: Laparoscopic Rectal Prolapse Surgery Study. An International, Double Cohort Study to Determine the Optimal Treatment for Rectal Prolapse.
Brief Title: An International Double Cohort Study to Compare Laparoscopic Ventral Rectopexy With Laparoscopic Resection Rectopexy
Acronym: LaProS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 2 patients enrolled lost of follow-up after completing 1st year visits.PI decided to close
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTR2743
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Rectal Prolapse; Procidentia
Keywords: Laparoscopic surgery; Colorectal Surgery; Quality of Life; Rectal Prolapse; Anorectal Physiology
MeSH Terms: conditions — Rectal Prolapse; Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 2 (Active Comparator): Cohort 2 (two) will consist of 120 patients with an external rectal prolapse (Oxford Grade V)treated by Laparoscopic Resection Rectopexy (LRR). These patients will be included in the US centers involved in this study and treated by LRR.
  Interventions: Procedure: Laparoscopic Resection Rectopexy
- Cohort 1 (Active Comparator): Cohort one will consist of 120 patients with an external rectal prolapse (Oxford Grade V) which will be treated with Laparoscopic Ventral Rectopexy. As this is the standard treatment in the European centers involved in this study these patients will be selected in the participating centers in the Netherlands, Belgium and England.
  Interventions: Procedure: Laparoscopic Ventral Rectopexy

INTERVENTIONS:
Procedure: Laparoscopic Resection Rectopexy — laparoscopic sigmoidectomy with suture rectopexy
  Other Names: Laparoscopic Resection Rectopexy,
  Arms: Cohort 2
Procedure: Laparoscopic Ventral Rectopexy — laparoscopic ventral rectopexy with mesh
  Other Names: Laparoscopic ventral mesh rectopexy; Ventral mesh rectopexy
  Arms: Cohort 1

SUMMARY:
Background:

Rectal prolapse (RP) is the descent of the upper rectum and is a common problem in the western world. Surgery is the only definite treatment and is preferably performed minimally invasive. High-level prospective studies on treatment strategies for RP currently are lacking and, thus, no consensus exist regarding the optimal treatment for patients with RP. Furthermore, remarkable transatlantic differences exist, as in Europe, laparoscopic ventral rectopexy (LVR) is regarded the treatment of choice, while in the USA Laparoscopic Resection Rectopexy (LRR) remains the golden standard.

Objective:

To determine the optimal minimally invasive surgical treatment for patients with RP.

Design:

International, prospective, comparative double cohort study. The first cohort will consist of 120 European patients with a RP and will be treated with LVR. Centres in The Netherlands, Belgium and the UK are enlisted for participation. The second cohort will consist of 120 American patients with a RP, treated with LRR. Several US centres are enlisted. Preoperative work-up consists of radiological imaging and standardised questionnaires. Follow-up (FU) is set on two years. During FU, pre-operative imaging and questionnaires will be repeated.

Primary & secondary outcomes:

Primary endpoint will be improvement on the Gastro-Intestinal-Quality-of-Life-Index (GIQLI). Secondary endpoints will be generic Quality-of-Life, functional results, morbidity, mortality, recurrences and cost-effectiveness.

Time frame:

Study and inclusion start will be on January the 1st, 2011 and will take approximately 18-24 months. Therefore, total study duration will be 42-48 months.

DETAILED DESCRIPTION:
A Rectal Prolapse (RP), or procidentia, is the descent of the upper rectum. This descensus in the full-thickness of the rectum, and can be either internal, called an internal rectal prolapse or intussusception (IRP), or through the anus (called an external rectal prolapse (ERP)).

RP mainly occurs in women (80-90%) of which most in the 6-7th decade. Risk factors for developing a rectal prolapse are the presence of an abnormal deep pouch of Douglas, laxity and atonic condition of the muscles of the pelvic floor and anal canal. Moreover, weakness of both internal and external sphincters, often with evidence of pudendal nerve neuropathy and the lack of normal fixation of the rectum may lead to RP. This also frequently leads to other pelvic organ prolapses like vesicoceles, enteroceles and genital prolapses. In this study the investigators will focus on the treatment of RP.

Rectal prolapses cause anal incontinence in more than half of the patients. Another frequent symptom of RP is constipation. Furthermore, the rectal prolapse can lead to anal pain as a result of incarceration leading to ulcers, necrosis and perforation.

Besides the fact that this disease has a considerable impact on the individual quality of life, it also carries significant socio-economic consequences as incontinence products have to be used in large amounts.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an indication for Laparoscopic Resection Rectopexy* for External Rectal Prolapse (Oxford Grade V)

Exclusion Criteria:

* Under 18 years of age
* Former rectosigmoid resection
* Former rectal prolapse surgery
* Rectosigmoid tumor
* Severe mental retardation
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 24 months
  Quality of Life objectified by the gastro-Intestinal Quality of Life Index and secondary by EuroQoL-5D and Short-Form 36 questionnaires.

SECONDARY OUTCOMES:
Optimal surgery and functional results | 24 months
  Compare 2 laparoscopic approaches and functional results evaluated by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Wexner, MD, Principal Investigator — Cleveland Clinic Floria
Locations (6):
- United States (6):
  - The Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Floria, Weston, Florida
  - Oschner Clinic North Shore, New Orleans, Louisiana
  - John Hopkins, Baltimore, Maryland
  - Lahey Medical Center, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: No